CLINICAL TRIAL: NCT00616837
Title: Remote Orthopedic Outpatient Consultation by Help of Telemedicine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: Helse Nord (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: P-REK-N-134/2006; Personvernombudet,UNN 05.12.06 (Other: University Hospital North Norway); P-REK-N-134/2006 (REK) (Registry Identifier: Regional ethic comittee, Region North)
Record Dates: First submitted 2008-01-22; First posted 2008-02-15 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Orthopedic Disorders
Keywords: Remote consultation/*methods; Orthopaedics methods; Telemedicine; Follow-up study; Ambulatory care
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard consultation (Active Comparator): Standard care in orthopaedic outpatient clinic
  Interventions: Other: Standard care in orthopaedic outpatient clinic
- Telemedicine consultation (Experimental): Orthopaedic care in outpatient clinic by use of telemedicine.
  Interventions: Other: Telemedicine consultation

INTERVENTIONS:
Other: Telemedicine consultation — Outpatient consultation by help of telemedicine (video conference)
  Arms: Telemedicine consultation
Other: Standard care in orthopaedic outpatient clinic — Standard care in orthopedic outpatient clinic (usual care)
  Arms: Standard consultation

SUMMARY:
Patients from 4 local communities in northern Norway referred (either new or follow up) to orthopaedic department, University hospital of Northern Norway for outpatient consultation, are randomly assigned to either remote consultation by use of telemedicine (camera and screen), or standard consultation at the hospital. There are x-ray facilities also at the remote site. The patients randomized to telemedicine consultation meet special trained nurses at the remote site, but doctor only by video conference. The patients will be followed for up to one year. The primary endpoint is quality of care achieved with the telemedicine consultation as compared to standard outpatient consultation (assessed by questionnaires filled out by the doctor involved). Secondary end points are patient satisfaction assessed by questionnaires and economic analyses. The study hypothesis is non-inferiority of telemedicine consultation vs. conventional, outpatient consultation.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent given
* New referred patients to orthopaedic department (outpatient), UNN, for conditions suitable for telemedicine consultation
* Follow up consultation of trauma patients (operated/not operated)
* Follow up consultation after elective orthopaedic surgery (e.g hip prothesis)
* Follow up of other orthopaedic patients

Exclusion Criteria:

* Senile dementia
* Soldiers, prisoners
* Patients not talking Norwegian, dependent on translator
* If specialized procedures are required during follow up (e.g. cat-scan, ultrasound etc)
* Patients requiring a specific doctor

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2007-11; Primary Completion 2012-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Safety and quality of health care | 1 year

SECONDARY OUTCOMES:
Patient satisfaction | up to 1 year after last consultation
  Patient satisfaction will be measured based on a total score calculated on the basis of responses to satisfaction questionnaire. Questionnaires will be filled out at each visit/consultation and at 3 months or one year after last consultation.
Cost value | up to 1 year
  Travel expenses, escort expenses, equipment and other costs related to patient consultation

CONTACTS AND LOCATIONS:
Overall Officials: Astrid S Buvik, MD, Principal Investigator — University Hospital North Norway; Arvid Smaabrekke, MD, Study Chair — University Hospital North Norway; Jan Abel Olsen, PhD, Study Chair — University of Tromso; Tom Wilsgaard, PhD, Study Director — University of Tromso, Norway; Gunnar Knutsen, MD, PhD, Study Chair — University Hospital NorthNorway
Locations (1):
- Orthopaedic department, Tromso University Hospital, Tromsø, Norway

REFERENCES:
- [Derived] Buvik A, Bergmo TS, Bugge E, Smaabrekke A, Wilsgaard T, Olsen JA. Cost-Effectiveness of Telemedicine in Remote Orthopedic Consultations: Randomized Controlled Trial. J Med Internet Res. 2019 Feb 19;21(2):e11330. doi: 10.2196/11330. PMID 30777845
- [Derived] Buvik A, Bugge E, Knutsen G, Smabrekke A, Wilsgaard T. Quality of care for remote orthopaedic consultations using telemedicine: a randomised controlled trial. BMC Health Serv Res. 2016 Sep 8;16(1):483. doi: 10.1186/s12913-016-1717-7. PMID 27608768